CLINICAL TRIAL: NCT01544491
Title: A 12-month, Multicenter, Open Label, Randomized, Controlled Study to Evaluate the Efficacy, Tolerability and Safety of Early Introduction of Everolimus, Reduced CNI, and Early Steroid Elimination Compared to Standard CNI, Mycophenolate Mofetil and Steroid Regimen in Paediatric Renal Transplant Recipients With a 24-month Additional Safety Follow-up.
Brief Title: Efficacy, Tolerability and Safety of Early Introduction of Everolimus, Reduced Calcineurin Inhibitors and Early Steroid Elimination Compared to Standard CNI, Mycophenolate Mofetil and Steroid Regimen in Paediatric Renal Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001A2314; 2010-024381-21 (EudraCT Number)
Record Dates: First submitted 2011-06-09; First posted 2012-03-06 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Prevention of Acute Rejection in Paediatric Recipients of a Renal Transplant
Keywords: Paediatric kidney transplantation; Early MMF to everolimus conversion; Composite efficacy (biopsy-proven acute rejection, graft loss or death); Renal function
MeSH Terms: conditions — Death | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Investigational arm (Experimental): Conversion from MMF to everolimus plus reduced dose tacrolimus and steroids withdrawal at 6 months after transplant
  Interventions: Drug: RAD001
- Control arm (Active Comparator): MMF continuation (in combination with tacrolimus and standard dose steroids)
  Interventions: Drug: MMF

INTERVENTIONS:
Drug: RAD001 — Everolimus (C0 trough level of 3-8 ng/mL) in combination with reduced dose tacrolimus and steroids withdrawal at 6 months after transplant
  Arms: Investigational arm
Drug: MMF — MMF (Cellcept®): 600mg/m2/dose twice daily (1200 mg/m2/day) in combination with tacrolimus (Prograf) and standard dose steroids
  Arms: Control arm

SUMMARY:
The purpose of this study is to determine if everolimus combined with reduced exposure CNI (TAC) is efficacious and safe and will support corticosteroid elimination compared to a standard exposure CNI (TAC) + MMF + steroid regimen after paediatric kidney transplantation. An additional purpose of the study is to assess the effect of the combination of EVR and reduced exposure CNI (TAC) on renal function.

This study is part of the requirements of the Paediatric Investigational Plan approved by Paediatric Committee at the European Medicines Agency (PDCO/EMA) on September 10, 2010, and is intended to support the indication of everolimus in the prevention of acute rejection in paediatric recipients of a renal transplant.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria at baseline:

1. Written informed consent/assent must be obtained from the parent(s) or legal guardian before any assessment is performed.
2. Primary or secondary paediatric kidney transplant recipient aged greater than or equal to 1 year and younger than 18 years receiving a deceased donor or non-HLA identical living donor (related or unrelated) renal transplant.

Inclusion criteria at randomization:

1. Patients on TAC + MMF + steroids.
2. Renal function with eGFR > 40 ml/min/1.73 m2 (Schwartz formula - abbreviated).

Exclusion Criteria:

Exclusion criteria at baseline:

1. Recipients of kidneys from donors with known renal disease (such as diabetes nephropathy, nephrosclerosis), at the time of transplant.
2. Recipients of a kidney with a cold ischemia time > 24 hours.
3. History of hypersensitivity or contraindications to any of the study drugs or to drugs of similar chemical classes, or to any of the excipients.
4. History of malignancy of any organ system treated or untreated, carrying possible risk of recurrence according to current guidelines (Appendix 10 of protocol).

Exclusion criteria at randomization:

1. Use of other investigational drugs at the time of randomization, or within 30 days or 5 half-lives prior randomization, whichever is longer.
2. Patients with ongoing or recently (within 2 weeks prior to randomization) treated episodes of acute rejection (any grade) or a steroid resistant acute rejection at the time of randomization.
3. Patients who experienced acute cellular rejection (Banff ≥1B) or any antibody mediated acute rejection or patients considered at high risk of antibody mediated acute rejection by the investigator assessment (e.g. presence of newly formed DSA, histological suspicion) at any time before randomization (as the DSA quantitative threshold to define high risk is not fully established, the assessment of the risk will be made after discussion between the laboratory expert and the investigator who will take into account all information available and apply best judgment).
4. Patients with ongoing wound healing problems, clinically significant wound infection requiring continued therapy or other severe surgical complication in the opinion of the investigator.
5. Patients who are treated with drugs that are strong inducers or inhibitors of cytochrome P450 3A4 (CYP3A4) and can not discontinue the treatment (see Appendix 6 for list of medications).
6. Patients with nephrotic range proteinuria (protein to creatinine ratio ≥2.0 mg/mg or 200 mg/mmol (Hogg, 2003).

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 106 (Actual)
Dates: Start 2012-08-17 (Actual); Primary Completion 2016-10-03 (Actual); Study Completion 2018-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (30):
- United States (3):
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, St Louis, Missouri
- Novartis Investigative Site, Santa Fe, Argentina
- Brazil (2):
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
- France (3):
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Paris
- Germany (7):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Tübingen
- Novartis Investigative Site, Budapest, Hungary
- Italy (5):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Roma, ITA
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Torino, TO
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Warsaw, Poland
- Novartis Investigative Site, Esplugues de Llobregat, Barcelona, Spain
- Novartis Investigative Site, Stockholm, Sweden
- Novartis Investigative Site, Antalya, Turkey (Türkiye)
- United Kingdom (3):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Nottingham

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Patry C, Sauer LD, Sander A, Krupka K, Fichtner A, Brezinski J, Geissbuhler Y, Aubrun E, Grinienko A, Strologo LD, Haffner D, Oh J, Grenda R, Pape L, Topaloglu R, Weber LT, Bouts A, Kim JJ, Prytula A, Konig J, Shenoy M, Hocker B, Tonshoff B. Emulation of the control cohort of a randomized controlled trial in pediatric kidney transplantation with Real-World Data from the CERTAIN Registry. Pediatr Nephrol. 2023 May;38(5):1621-1632. doi: 10.1007/s00467-022-05777-x. Epub 2022 Oct 20. PMID 36264431
- [Derived] Tonshoff B, Tedesco-Silva H, Ettenger R, Christian M, Bjerre A, Dello Strologo L, Marks SD, Pape L, Veldandi U, Lopez P, Cousin M, Pandey P, Meier M. Three-year outcomes from the CRADLE study in de novo pediatric kidney transplant recipients receiving everolimus with reduced tacrolimus and early steroid withdrawal. Am J Transplant. 2021 Jan;21(1):123-137. doi: 10.1111/ajt.16005. Epub 2020 Jun 27. PMID 32406111

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Full Analysis set (FAS) 106 enrolled and randomized patients except misrandomized Per Protocol set (PPS) 90 patients in the FAS without major protocol deviations Safety set (SAF) 106 randomized patients who received at least one dose of study drug
Groups:
- EVR+rTAC: Investigational arm : Conversion from MMF to everolimus plus reduced dose tacrolimus and steroids withdrawal at 6 months after transplant
- MMF+sTAC: Control arm : MMF continuation (in combination with tacrolimus and standard dose steroids)
Period: Overall Study
Arm/Group | EVR+rTAC | MMF+sTAC
Started | 52 | 54
Completed | 47 | 51
Not Completed | 5 | 3
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — administrative problems | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EVR+rTAC | MMF+sTAC | Total
Number analyzed (Participants) | 52 | 54 | 106
Age, Customized [Count of Participants; unit: Participants]
  1 to <11 years | 26 | 27 | 53
  11 <= 18 years | 26 | 27 | 53
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 29 | 31 | 60
  Female | 23 | 23 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 42 | 47 | 89
  Black | 1 | 0 | 1
  Asian | 3 | 2 | 5
  Other | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Having Reached the Composite Efficacy Endpoint of Biopsy-proven Acute Rejection
Description: To estimate the rate of the composite efficacy endpoint of biopsy-proven acute rejection (BPAR), graft loss or death at 12 months post transplantation in primary paediatric kidney transplant recipients converted at 4-6 weeks post-transplantation from MMF + standard TAC regimen and steroids, to everolimus + reduced dose TAC regimen and steroid withdrawal at 6 months, versus continuation of MMF + standard TAC regimen and steroids.
Time Frame: 12 months, 36 months
Population: Full Analysis set (12 months and 36 months) Results given as number of participants with composite efficacy failures
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+rTAC | MMF+sTAC
Number analyzed (Participants) | 52 | 54
Participants
  12 months | 5 | 3
  36 months | 5 | 5
Statistical Analysis 1: Comparison: EVR+rTAC vs MMF+sTAC; at 12 months; Test type: Non-Inferiority — Kaplan-Meier estimates and between treatment differences are estimated using the Kaplan-Meier product-limit formula and 80% confidence intervals derived using standard errors estimated from Greenwood's formula; p = 0.9712, Log Rank; Mean Difference (Final Values) = 0.1, 80% CI 2-sided [-6.6 to 6.8], Standard Error of Mean 5.25
Statistical Analysis 2: Comparison: EVR+rTAC vs MMF+sTAC; 36 months; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.9634, Log Rank; Mean Difference (Final Values) = 0.2, 80% CI 2-sided [-7.3 to 7.7], Standard Error of Mean 5.84

2. Primary Outcome: To Evaluate Renal Function, Assessed by Glomerular Filtration Rate (eGFR) and Estimated by the Schwartz Formula (Abbreviated), at Month 12 and 36
Description: To evaluate renal function assessed by Glomerular Filtration Rate (eGFR) estimated by the Schwartz Formula (abbreviated) (Schwartz, 2009).
Time Frame: 12 months and 36 months post-transplantation
Population: Full Analysis set 12 months and 36 months
Measure: Mean (Standard Error); unit: mL/min/1.73m2
Arm/Group | EVR+rTAC | MMF+sTAC
Number analyzed (Participants) | 52 | 54
mL/min/1.73m2
  12 months: number analyzed (Participants) | 44 | 48
  12 months | 76.7 (3.66) | 71.7 (3.56)
  36 months | 68.1 (3.45) | 67.3 (3.54)
Statistical Analysis 1: Comparison: EVR+rTAC vs MMF+sTAC; at 12 months; Test type: Non-Inferiority — KM estimates and between treatment differences are estimated using the Kaplan-Meier product-limit formula and 80% confidence intervals derived using standard errors estimated from Greenwood's formula; p = 0.3455, t-test, 2 sided; Mean Difference (Net) = 5.0, 80% CI 2-sided [-1.8 to 11.8], Standard Error of Mean 5.26
Statistical Analysis 2: Comparison: EVR+rTAC vs MMF+sTAC; 36 months; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p = 0.8642, t-test, 2 sided; Mean Difference (Final Values) = 0.8, 80% CI 2-sided [-5.5 to 7.2], Standard Error of Mean 4.95

3. Secondary Outcome: Composite Efficacy Endpoint
Description: To evaluate the proportion of patients with the following efficacy events: Biopsy Proven Acute Rejection (BPAR), graft loss or death. The efficacy events will be descriptively summarized by treatment group.
Time Frame: at 12 and 36 months post-transplantation
Population: full Analysis set 36 month analysis Results given as number of participants with composite efficacy failures
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+rTAC | MMF+sTAC
Number analyzed (Participants) | 52 | 54
Participants
  month 12 composite efficacy endpoint | 5 | 3
  graft loss 12 months | 0 | 0
  death 12 months | 0 | 0
  acute rejection 12 months | 5 | 4
  treated acute rejection 12 months | 5 | 4
  Biopsy proven acute rejection 12 months | 5 | 3
  treated Biopsy proven acute rejection 12 months | 5 | 3
  month 36 composite efficacy endpoint | 5 | 5
  graft loss 36 months | 1 | 2
  death 36 months | 0 | 0
  acute rejection 36 months | 5 | 7
  Biopsy proven acute rejection 36 months | 5 | 5
  treated Biopsy proven acute rejection 36 months | 5 | 5

4. Secondary Outcome: To Evaluate the Severity of BPAR (Acute T-cell Mediated Rejection Only) (Banff 2009)
Description: T-cell mediated rejection severity :
  Type IA - Significant interstitial infiltration (> 25% of parenchyma) and foci of moderate tubulitis (> 4 mononuclear cells/tubular cross section or group of 10 tubular cells).
  Type IB - Significant interstitial infiltration (> 25% of parenchyma) and foci of severe tubulitis (> 10 mononuclear cells/tubular cross section or group of 10 tubular cells).
  Type IIA - Mild to moderate intimal arteritis Type IIB - Severe intimal arteritis comprising > 25% of the lumenal area Type III - Transmural (full vessel wall thickness) arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells (with accompanying lymphocytic inflammation)
Time Frame: month 12, month 36
Population: full Analysis set 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+rTAC | MMF+sTAC
Number analyzed (Participants) | 52 | 54
Participants
  month 12 grade IA | 3 | 1
  month 12 grade IB | 1 | 0
  month 12 grade IIA | 0 | 2
  month 12 grade IIB | 0 | 0
  month 12 grade III | 0 | 0
  month 36 grade IA | 3 | 1
  month 36 grade IB | 2 | 0
  month 36 grade IIA | 0 | 1
  month 36 grade IIB | 0 | 1
  month 36 grade III | 0 | 1

5. Secondary Outcome: To Evaluate the Time to Event of BPAR
Description: Time to incidence of Event, given in terms of number of participants with an Event according to time interval up to 36 months
Time Frame: 36 months
Population: full Analysis set, 36 month analysis
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+rTAC | MMF+sTAC
Number analyzed (Participants) | 52 | 54
Participants
  day 1-7 | 0 | 0
  day 8-14 | 0 | 0
  day 15-28 | 1 | 0
  day 29-56 | 0 | 0
  day 57-84 | 0 | 0
  day 85-150 | 2 | 2
  day 151- 240 | 0 | 0
  day 241-330 | 1 | 2
  day 331- 510 | 0 | 1
  day 511-690 | 1 | 0
  day 691-870 | 0 | 0
  day 871-1050 | 0 | 0
  after day 1050 | 0 | 0

6. Secondary Outcome: Incidence of Biopsy Proven Antibody Mediated Rejection.
Description: To evaluate the proportion of patients with the following efficacy events: biopsy proven antibody mediated rejection/Steroid resistant BPAR and BPAR treated with T cell depleting therapy.
Time Frame: at 12 and 36 months post-transplantation
Population: Full Analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+rTAC | MMF+sTAC
Number analyzed (Participants) | 52 | 54
Participants
  patients with BPAR at 12 months | 7 | 8
  BPAR Steroid resistant,12 months | 1 | 0
  BPAR, T Cell depleting therapy 12 months | 1 | 1
  patients with BPAR at 36 months | 6 | 12
  BPAR Steroid resistant,36 months | 1 | 2
  BPAR, T Cell depleting therapy 36 months | 2 | 1

7. Secondary Outcome: Chronic Allograft Nephropathy / Interstitial Fibrosis and Tubular Atrophy
Description: To evaluate the proportion of patients with chronic allograft nephropathy (interstitial fibrosis and tubular atrophy, IF/TA) by histopathology and its progression.The term chronic allograft nephropathy was used inappropriately in the protocol and therefore, replaced by interstitial fibrosis and tubular atrophy
Time Frame: at 12 and 36 months post-transplantation.
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+rTAC | MMF+sTAC
Number analyzed (Participants) | 52 | 54
Participants
  12 months | 3 | 3
  36 months | 11 | 7

8. Secondary Outcome: Proteinuria (Urinary Protein/Creatinine Ratio)
Description: The urinary protein/creatinine ratio will be descriptively summarized by treatment group at each visit. The incidence rate of patients with proteinuria will be categorized in <0.2 g/mg/mg, 0.2<2.0 mg/mg and ≥ 2.0 mg/mg and summarized by treatment groups at each visit.
Time Frame: at 12 and 36 months post-transplantation
Population: full analysis set 36 months analysis
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+rTAC | MMF+sTAC
Number analyzed (Participants) | 52 | 54
Participants
  Baseline < 200mg/g: number analyzed (Participants) | 27 | 29
  Baseline < 200mg/g | 1 | 2
  Baseline 200 - < 2000 mg/g: number analyzed (Participants) | 27 | 29
  Baseline 200 - < 2000 mg/g | 12 | 12
  Baseline >= 2000 mg/g: number analyzed (Participants) | 27 | 29
  Baseline >= 2000 mg/g | 14 | 15
  Month 12 < 200mg/g: number analyzed (Participants) | 32 | 39
  Month 12 < 200mg/g | 19 | 28
  Month 12 200 - < 2000 mg/g: number analyzed (Participants) | 32 | 39
  Month 12 200 - < 2000 mg/g | 13 | 11
  Month 12 >= 2000 mg/g: number analyzed (Participants) | 32 | 39
  Month 12 >= 2000 mg/g | 0 | 0
  Month 36 < 200mg/g: number analyzed (Participants) | 34 | 34
  Month 36 < 200mg/g | 23 | 23
  Month 36 200 - < 2000 mg/g: number analyzed (Participants) | 34 | 34
  Month 36 200 - < 2000 mg/g | 10 | 11
  Month 36 >= 2000 mg/g: number analyzed (Participants) | 34 | 34
  Month 36 >= 2000 mg/g | 1 | 0

9. Secondary Outcome: Growth/Development : Weight, Height, BMI : Change From Baseline
Description: Evaluation of the potential effects upon the bone growth. The Z-score is a statistical tool which helps to assess data (here child growth parameters) relative to a reference or standard population. The Z-score describes the distance and direction of an observation away from the population median (or mean, however, here the median was used). A negative Z-score shows that data are lower than the median of the standard population, a positive Z-score shows that data are higher than the median of the standard population, and a Z-score of zero shows that the data are equal to the median of the standard population. The more the Z-score is distant from 0, the more expressed is for example underweight or overweight.
Time Frame: month 12 , month 36 post transplantation.
Population: safety set, 36 months analysis
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | EVR+rTAC | MMF+sTAC
Number analyzed (Participants) | 52 | 54
z score
  Height month 12: number analyzed (Participants) | 37 | 48
  Height month 12 | 0.37 (0.625) | 0.20 (0.537)
  Height month 36: number analyzed (Participants) | 31 | 40
  Height month 36 | 0.72 (1.131) | 0.39 (0.776)
  Weight month 12: number analyzed (Participants) | 37 | 48
  Weight month 12 | 0.30 (0.732) | 0.42 (0.747)
  Weight month 36: number analyzed (Participants) | 31 | 40
  Weight month 36 | 0.61 (0.987) | 0.82 (1.268)
  BMI month 12: number analyzed (Participants) | 37 | 48
  BMI month 12 | 0.00 (0.716) | 0.24 (0.980)
  BMI month 36: number analyzed (Participants) | 31 | 40
  BMI month 36 | 0.02 (0.860) | 0.47 (1.231)

10. Secondary Outcome: Evaluation of Evolution of Renal Allograft Function Over Time
Description: results given as eGFR values by time interval
Time Frame: baseline, 6 months, 12 months , 24 months, 36 months
Population: full Analysis set 36 months
Measure: Mean (Standard Deviation); unit: ml/min/1.73m2
Arm/Group | EVR+rTAC | MMF+sTAC
Number analyzed (Participants) | 52 | 54
ml/min/1.73m2
  baseline: number analyzed (Participants) | 33 | 41
  baseline | 14.2 (11.38) | 13.1 (15.62)
  month 6: number analyzed (Participants) | 37 | 39
  month 6 | 76.6 (28.29) | 68.3 (21.02)
  month 12: number analyzed (Participants) | 32 | 42
  month 12 | 76.9 (21.61) | 67.8 (23.57)
  month 24: number analyzed (Participants) | 34 | 40
  month 24 | 72.9 (28.43) | 68.6 (23.26)
  month 36: number analyzed (Participants) | 34 | 35
  month 36 | 68.2 (21.60) | 69.6 (20.01)

11. Secondary Outcome: To Evaluate Renal Function, Assessed by Glomerular Filtration Rate (eGFR) and Estimated by the Schwartz Formula (Extended), at Month 12
Description: To evaluate renal function assessed by Glomerular Filtration Rate (eGFR) estimated by the Schwartz Formula (extended) (Schwartz, 2009). Results given as change from randomization
Time Frame: 12 months post-transplantation
Population: Full Analysis set 12 months months
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Arm/Group | EVR+rTAC | MMF+sTAC
Number analyzed (Participants) | 52 | 54
mL/min/1.73m2 | 4.6 (11.94) | -0.0 (23.92)

ADVERSE EVENTS:
Time Frame: up to 36 months
Description: AE additional description
Groups:
- EVR+rTAC: EVR+rTAC
- MMF+sTAC: MMF+sTAC
Arm/Group | EVR+rTAC | MMF+sTAC
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/54
Other Adverse Events (participants affected / at risk) | 46/52 | 48/54
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EVR+rTAC (N=52) | MMF+sTAC (N=54)
Anaemia (Blood and lymphatic system disorders) | 10 | 11
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 6 | 6
Neutropenia (Blood and lymphatic system disorders) | 2 | 10
Polycythaemia (Blood and lymphatic system disorders) | 3 | 0
Ear pain (Ear and labyrinth disorders) | 5 | 5
Abdominal pain (Gastrointestinal disorders) | 7 | 6
Abdominal pain upper (Gastrointestinal disorders) | 6 | 5
Aphthous ulcer (Gastrointestinal disorders) | 9 | 1
Constipation (Gastrointestinal disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 13 | 16
Mouth ulceration (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 4 | 4
Vomiting (Gastrointestinal disorders) | 10 | 8
Fatigue (General disorders) | 3 | 2
Pain (General disorders) | 3 | 3
Pyrexia (General disorders) | 14 | 11
BK virus infection (Infections and infestations) | 4 | 8
Bronchitis (Infections and infestations) | 2 | 4
Cystitis (Infections and infestations) | 3 | 1
Cytomegalovirus infection (Infections and infestations) | 3 | 3
Cytomegalovirus viraemia (Infections and infestations) | 0 | 3
Ear infection (Infections and infestations) | 1 | 5
Epstein-Barr viraemia (Infections and infestations) | 3 | 2
Epstein-Barr virus infection (Infections and infestations) | 7 | 2
Gastroenteritis (Infections and infestations) | 4 | 5
Influenza (Infections and infestations) | 3 | 1
Nasopharyngitis (Infections and infestations) | 16 | 6
Oral herpes (Infections and infestations) | 2 | 3
Otitis media (Infections and infestations) | 4 | 1
Pharyngitis (Infections and infestations) | 6 | 1
Rhinitis (Infections and infestations) | 7 | 5
Sinusitis (Infections and infestations) | 1 | 3
Tonsillitis (Infections and infestations) | 3 | 8
Upper respiratory tract infection (Infections and infestations) | 8 | 6
Urinary tract infection (Infections and infestations) | 13 | 15
Blood creatinine increased (Investigations) | 3 | 6
Hepatic enzyme increased (Investigations) | 3 | 1
Weight decreased (Investigations) | 0 | 5
Weight increased (Investigations) | 5 | 2
Acidosis (Metabolism and nutrition disorders) | 1 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 4
Iron deficiency (Metabolism and nutrition disorders) | 6 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 3 | 0
Obesity (Metabolism and nutrition disorders) | 2 | 3
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Headache (Nervous system disorders) | 10 | 11
Tremor (Nervous system disorders) | 1 | 4
Haematuria (Renal and urinary disorders) | 3 | 3
Proteinuria (Renal and urinary disorders) | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 5 | 2
Hypertension (Vascular disorders) | 7 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.